CLINICAL TRIAL: NCT07177404
Title: Surveying Experiences and Lifestyle Effects in Choosing Technology and Hybrid Closed Loop in Type 1 Diabetes
Brief Title: Choices and Experiences Around Closed-loop Therapy in Type 1 Diabetes
Acronym: SELECT HCL
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 25026
Record Dates: First submitted 2025-09-01; First posted 2025-09-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabete Mellitus; Type 1 Diabetes Mellitus
Keywords: Diabetes mellitus; Type 1 Diabetes Mellitus; Hybrid Closed Loop; Automated Insulin Delivery; Patient survey; Survey
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Type 1 diabetes requires a lot of work to try to keep glucose levels in the target range. Hybrid closed- loop, also known as artificial pancreas, takes glucose readings from a sensor (continuous glucose monitor) and uses an algorithm to tell an insulin pump how much insulin to deliver. Hybrid closed-loop has currently been rolled out to many people with type 1 diabetes in England. We are keen to develop a deeper understanding of the perspective of people living with type 1 diabetes who have choices about which hybrid closed-loop systems fit their needs.

The main purpose of this study is to explore the choices and experiences of people living with type 1 diabetes regarding closed-loop therapy.

DETAILED DESCRIPTION:
This is a cross-sectional online survey study, which involves people with type 1 diabetes who use closed-loop, wait to start closed-loop or considering closed-loop.

The primary objective of the study is to explore the factors driving the choices of people living with type 1 diabetes regarding closed-loop therapy.

The secondary objectives of the study are:

* To understand what treatment satisfaction with closed-loop therapy means to people living with type 1 diabetes
* To understand what additional support is needed for people with type 1 diabetes using closed-loop therapy

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years (no upper age limit)
* Type 1 diabetes (any duration)
* People who use closed-loop therapy or wait to start closed-loop therapy or considering closed-loop therapy in the future
* Ability to give informed consent

Exclusion Criteria:

* Any other type of diabetes apart from type 1 diabetes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be approached via their usual University Hospitals of Derby & Burton NHS diabetes care team.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ranking of factors influencing the choice of closed-loop therapy among people with type 1 diabetes | Day 1

SECONDARY OUTCOMES:
Ranking of factors contributing to treatment satisfaction with closed-loop therapy | Day 1
Distribution of responses to 5-point Likert scale questions assessing factors contributing to treatment satisfaction with closed-loop therapy | Day 1
Distribution of responses to 5-point Likert scale questions assessing the support needs of people using closed-loop therapy | Day 1
Associations of demographics and reported glucose levels with factors influencing the choice of closed-loop therapy | Day 1
Associations of demographics and reported glucose levels with factors contributing to treatment satisfaction with closed-loop therapy | Day 1
Associations of demographics and reported glucose levels with support needs related to closed-loop therapy | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby and Burton, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No